CLINICAL TRIAL: NCT02180880
Title: Symptom-Based Treatment for Neuropathic Pain in Spinal Cord Injured Patients, Randomized Clinical Trial
Brief Title: Symptom Based Treatment of Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ju Seok Ryu (Other)
Responsible Party: Sponsor-Investigator, Ju Seok Ryu, Assistant professor, CHA University
Organization: CHA University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuropathicPain
Record Dates: First submitted 2014-06-05; First posted 2014-07-03 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Neuralgia; Spinal Cord Injury
Keywords: Neuralgia; Spinal cord; Oxcarbazepine; Pregabalin; Drug therapy; Algorithms
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries | interventions — Pregabalin; Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregabalin and Oxcarbazpepine (Experimental): Pregabalin and Oxcarbazepine
  Interventions: Drug: Pregabalin and Oxcarbazepine

INTERVENTIONS:
Drug: Pregabalin and Oxcarbazepine — Subjects will take pregabalin for the duration of 2 weeks. The dosage will be increased from 75 mg twice to 150 mg twice a day.
  Subjects will stop pregabalin for 1 week and take oxcarbazepine 150mg twice.
  Other Names: Lyrica and Oxcarb

SUMMARY:
1. Neuropathic pain in spinal cord injured patients

1. Inclusion criteria

   * pain intensity, visual analogue scale > 3
   * a LANSS (Leeds assessment of neuropathic symptoms and signs) score of 12 and above
   * aged ≥20
2. Method

   * Stop pain medications
   * Test oxcarbazepine (150mg twice daily) and pregabalin (150mg twice daily)
   * Check pain intensity (VAS score) with Baron's classification

DETAILED DESCRIPTION:
In the present study, pharmacologic treatment included pregabalin and oxcarbazepine.

Stop medications such as Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), tramadol and anti-spastic drugs (baclofen, tizanidine) and other medications known to have effect on pain and the central nervous system prior to the study for at least 3 days.

1. Pain intensity (VAS score)

   1. 4 spontaneous characters

      * electric
      * burning
      * pricking
      * numbness
   2. evoked pain

      * allodynia
      * heat hyperalgesia
      * pressure hyperalgesia
2. Location of neuropathic pain

   1. neuropathic pain at level of spinal cord injury
   2. neuropathic pain below level of spinal cord injury

2. Side effects

ELIGIBILITY:
Inclusion Criteria:

* aged than 20 years
* Neuropathic pain symptoms : LANSS (Leeds assessment of neuropathic symptoms and signs) score of 12 and above
* Visual analogue scale score of 3 and above

Exclusion Criteria:

* No pregnancy
* systemic disease
* psychiatric disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Symptom based treatment of neuropathic pain | 2 week later
  Pain intensity using Visual analogue scale (0~100)

CONTACTS AND LOCATIONS:
Overall Officials: Ju Seok Ryu, MD, Study Chair — CHA University
Locations (1):
- CHA University, Seongnam-si, Kyounggi-do, South Korea

REFERENCES:
- [Derived] Min K, Oh Y, Lee SH, Ryu JS. Symptom-Based Treatment of Neuropathic Pain in Spinal Cord-Injured Patients: A Randomized Crossover Clinical Trial. Am J Phys Med Rehabil. 2016 May;95(5):330-8. doi: 10.1097/PHM.0000000000000382. PMID 26368836